CLINICAL TRIAL: NCT05369169
Title: Afferent Neurocardiac Signals, Cue Reactivity, and Cognitive Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Brandon Alderman, Ph.D., Associate Professor and Chair, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2021001073
Record Dates: First submitted 2022-03-16; First posted 2022-05-11 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Binge Drinking
Keywords: Alcohol Consumption; Baroreflex; Arousal; Breathing; Cardiovascular System; Cognition; Electrophysiology; Event-Related Potentials; Heavy Drinking; Attention; Individual Differences; Alcohol Cue; Brief Intervention; Cognitive Control; Cue Reactivity; Drinking Behavior; Young Adult; Heart Rate Variability
MeSH Terms: conditions — Binge Drinking; Alcohol Drinking; Respiratory Aspiration; Drinking Behavior

STUDY DESIGN:
Intervention Model Description: Subjects will complete an active treatment of slow resonance paced breathing and a control visual color block task on separate days, separated by approximately one week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resonance paced breathing (Experimental): Active resonance breathing task consisting of synchronizing breathing with a visual pacer (E-Z Air, Thought Technology, Ltd., Plattsburgh, NY) that moves up (inhale) and down (exhale) at the rate of 0.1 Hz (6 breaths per min)
  Interventions: Behavioral: Resonance breathing
- Low demand vanilla control (Active Comparator): A low-demand cognitive "vanilla" task wherein different colored rectangles are presented for 10 sec each, and participants are instructed to silently count the number of blue rectangles
  Interventions: Behavioral: Low demand cognitive task

INTERVENTIONS:
Behavioral: Resonance breathing — Participants will synchronize their breathing with a visual pacer (E-Z Air, Thought Technology, Ltd., Plattsburgh, NY) that moves up (inhale) and down (exhale) at the rate of 0.1 Hz (6 breaths per min)
  Arms: Resonance paced breathing
Behavioral: Low demand cognitive task — Different colored rectangles are presented for 10 sec each, and participants are instructed to silently count the number of blue rectangles
  Arms: Low demand vanilla control

SUMMARY:
Conscious attempts to regulate alcohol use are often undermined by automatic attention and arousal processes activated by alcohol cues, as well as by diminished ability to inhibit in-the-moment behaviors. The current study will examine whether a brief behavioral intervention of slow breathing paced at a resonance frequency of the cardiovascular system can interrupt automatic alcohol cue reactivity and enhance cognitive control in binge drinkers. Results from the proposed study may provide new prevention and intervention targets to interrupt unhealthy drinking behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Must report at least 2 binge drinking episodes in the past month
* Have normal or corrected-to-normal vision

Exclusion Criteria:

* History or presence of serious psychiatric disorders, neurological disorders, or head injury resulting in a loss of consciousness
* Presence of any serious medical condition
* Report of more than a few occasions (3-4) of illicit drug use, except for cannabis, in the preceding year

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants will self-identify gender identity on an approved demographic questionnaire
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
N2 ERP amplitude (in microvolts) elicited from an Alcohol Cued Go/No-Go task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  The N2 component (in microvolts) of the event-related potential occurring 250-350 ms after stimulus presentation at frontal and central electrode sites during an Alcohol Cued Go/No-Go task following a 5-minute course of resonance breathing compared to a low-demand control task
N2pc ERP amplitude (in microvolts) elicited from a visual dot probe detection task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  The N2pc component of the event-related potential occurring 200-275 ms after stimulus presentation at parietal and occipital electrode sites (ipsilateral minus contralateral hemisphere activity) during a modified visual dot probe detection task following a 5-minute course of resonance breathing compared to a low-demand control task
P3b ERP amplitude (in microvolts) elicited from a picture-viewing task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  The P3b component of the event-related potential occurring 300-600 ms after stimulus presentation at central and parietal electrode sites during a picture viewing task following a 5-minute course of resonance breathing compared to a low-demand control task
N2 ERP latency (in milliseconds) elicited from an Alcohol Cued Go/No-Go task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  The latency of the N2 component of the event-related potential from frontal and central electrode sites during a picture viewing task following a 5-minute course of resonance breathing compared to a low-demand control task. Latency will be determined using 50% area latency from a difference wave between task conditions
N2pc ERP latency (in milliseconds) elicited from a visual dot probe detection task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  The latency of the N2pc component of the event-related potential from parietal and occipital electrode sites during a visual dot probe detection task following a 5-minute course of resonance breathing compared to a low-demand control task. Latency will be determined using 50% area latency from a difference wave between task conditions
P3b ERP latency (in milliseconds) elicited from a picture-viewing task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  The latency of the P3b component of the event-related potential from central and parietal electrode sites during a picture viewing task following a 5-minute course of resonance breathing compared to a low-demand control task. Latency will be determined using 50% area latency from a difference wave between task conditions
Task accuracy from the behavioral response during the Alcohol Cued Go/No-Go task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  Task accuracy as a percentage of correct behavioral responses to the task during the Alcohol Cued Go/No-Go ERP task following a 5-minute course of resonance breathing compared to a low-demand control task
Reaction time from the behavioral response during the Alcohol Cued Go/No-Go task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  Reaction time for the correct behavioral responses to the task measured in milliseconds during the Alcohol Cued Go/No-Go ERP task following a 5-minute course of resonance breathing compared to a low-demand control task
Task accuracy from the behavioral response during the visual dot probe detection task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  Task accuracy as a percentage of correct behavioral responses to the task during the visual dot probe detection task following a 5-minute course of resonance breathing compared to a low-demand control task
Reaction time from the behavioral response during the visual dot probe detection task | Immediate; Difference between the active resonance breathing compared to the low demand cognitive task occurring one week apart
  Reaction time for the correct behavioral responses to the task measured in milliseconds during the visual dot probe ERP task following a 5-minute course of resonance breathing compared to a low-demand control task

CONTACTS AND LOCATIONS:
Overall Officials: Brandon L Alderman, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey; Marsha E Bates, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data via the NIAAA Data Archive (NIAAADA) repository within the larger National Institute of Mental Health (NIMH) Data Archive (NDA).
  Data generated by the proposed project include the following information on participants (male and female) aged 18-35 years:
  Surveys:
  * Basic Demographics (Age, Sex, Race/Ethnicity, Height/Weight)
  * Current Alcohol and Substance Use
  * Alcohol Use Questionnaire (AUQ), Penn Alcohol Craving Scale (PACS), and Alcohol Sensitivity Questionnaire
  Electrophysiological Data:
  * N2pc, P3b, and N2 components of the human event-related brain potential (ERP)
  * Collected during three cognitive tasks of cue reactivity (2) and inhibitory control (1)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the conclusion of data collection and no later than 24 months after the NIH award end date or 6 months post-publication of the final data set (whichever date occurs first). There is no restriction for how long the data will be available.